CLINICAL TRIAL: NCT01553240
Title: Neurocircuitry of Autism- fMRI and Transcranial Magnetic Stimulation Studies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator (Dr. Sporn) left the sponsoring institution.
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5438
Record Dates: First submitted 2011-07-19; First posted 2012-03-14 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Autism Spectrum Disorder; Asperger Disorder; Pervasive Developmental Disorder
Keywords: TMS; functional MRI; Supplementary motor cortex; Right Temporoparietal junction( RTPJ)
MeSH Terms: conditions — Autism Spectrum Disorder; Asperger Syndrome; Child Development Disorders, Pervasive | interventions — Transcranial Magnetic Stimulation; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TMS and fMRI (Experimental): * functional MRI
  * single and paired pulse TMS (to identify the difference of motor excitability between patients and healthy controls)
  Interventions: Device: TMS and functional MRI (Magstim)

INTERVENTIONS:
Device: TMS and functional MRI (Magstim) — single and paired pulse low frequency TMS. 3T structural MRI scans, amplitude modulated continuous arterial spin labeling( CASL) perfusion imaging sequence optimized for 3T is employed for perfusion MR scans using GE FAIR sequence for parallel imaging.
  Other Names: Magstim, Magstim 200, BISTIM Module

SUMMARY:
This study uses functional brain imaging and noninvasive brain stimulation techniques to study the brain basis of developmental disorders like Autism Spectrum Disorder and Asperger Disorder. Functional magnetic resonance imaging (fMRI) and recently approved FDA treatment of depression, Transcranial magnetic stimulation (TMS) will be used to study the neurocircuitry of certain symptom clusters in developmental disorders.

DETAILED DESCRIPTION:
The purpose of this research is to study areas of the brain that may have something to do with repetitive movements (things that people do over and over again) and difficulty communicating with other people (problems with talking to, understanding, or just being in a relationships with other people). The investigators are trying to find out why these brain areas are working differently in people with developmental disorders, such as Autism and how the investigators can one day improve them with new brain stimulation techniques.

The investigators will do screening to make sure that you are eligible for the study. After screening, the investigators will do functional MRI. In this procedure the subject or the control will be looking at videos developed to understand their social communication and language skills. The investigators will be able to understand differences of brain activation between patients and control. The investigators will also use TMS to identify the difference of motor excitability between patients and healthy control.

ELIGIBILITY:
Inclusion Criteria:

* for Healthy volunteer:

  * no current psychiatric disorder meeting Axis 1 DSM-4 criteria.
  * English speaking,
  * verbal and full scale IQ > 65,
  * capacity to give consent and signed HIPPA authorization.
* for Autism Spectrum Disorders:

  * diagnosed with Autism, Asperger or Pervasive Developmental Disorder not otherwise specified,
  * English speaking,
  * capacity to give consent and verbal and full scale IQ > 65,
  * signed HIPPA authorization,
  * participants currently taking psychotropic medications must be at the same stable doses and be willing to continue at the same dose through out the study

Exclusion Criteria:

* for Healthy control and ASD:

  * women of child bearing potential not using birth control pills or breast feeding,
  * h/o bipolar disorder (lifetime),
  * any psychotic disorder( lifetime),
  * history of major depressive disorder or of substance abuse or dependence within the past year,
  * verbal or full scale IQ less than or equal to 65,
  * intracranial implants,
  * metallic implants,
  * shrapnel in the body,
  * metallic braces,
  * cardiac pacemakers or
  * vagus nerve stimulation device,
  * claustrophobia,
  * prior dx of seizure,
  * increased intracranial pressure or history of significant head trauma with loss of consciousness for at least 5 minutes
  * current significant laboratory abnormality,
  * neurological disorder including but not limited to space occupying brain lesion,
  * any history of seizures,
  * history of cerebrovascular accidents,
  * fainting,
  * cerebral aneurysm,
  * dementia,
  * huntington,
  * chorea,
  * multiple sclerosis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2007-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Sporn, MD, Principal Investigator — NYPI, Columbia University; Sarah Lisanby, MD, Study Chair — NYPI, Columbia University
Locations (1):
- New York state Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Result] Bodfish JW, Symons FJ, Parker DE, Lewis MH. Varieties of repetitive behavior in autism: comparisons to mental retardation. J Autism Dev Disord. 2000 Jun;30(3):237-43. doi: 10.1023/a:1005596502855. PMID 11055459
- [Result] Baron-Cohen S, Wheelwright S, Skinner R, Martin J, Clubley E. The autism-spectrum quotient (AQ): evidence from Asperger syndrome/high-functioning autism, males and females, scientists and mathematicians. J Autism Dev Disord. 2001 Feb;31(1):5-17. doi: 10.1023/a:1005653411471. PMID 11439754
- [Result] Roid, G.H. Stanford Binet Intelligence Scles, Fifth Edition ( Riverside Publishing, Itasca, IL, 2003)
- [Result] Lord C, Rutter M, Le Couteur A. Autism Diagnostic Interview-Revised: a revised version of a diagnostic interview for caregivers of individuals with possible pervasive developmental disorders. J Autism Dev Disord. 1994 Oct;24(5):659-85. doi: 10.1007/BF02172145. PMID 7814313
- [Result] Lord C, Risi S, Lambrecht L, Cook EH Jr, Leventhal BL, DiLavore PC, Pickles A, Rutter M. The autism diagnostic observation schedule-generic: a standard measure of social and communication deficits associated with the spectrum of autism. J Autism Dev Disord. 2000 Jun;30(3):205-23. PMID 11055457
- [Result] APA. Diagnostic and Statistical Manual of Mental States Disorders. 4th ed. DSM-4-R( American Psychiatric Association, Washington, DC,2000)
- [Result] Sparrow, S., Cicchetti, D. & Balla,D. The Vineland-2 Adaptive Behavior Scales( Survey Interview Form) ( American Guidance Service, Circle Pines, MN, 2005)
- [Result] Constantino, J.N. The Social responsiveness Scale. ( Western psychological Services, Los Angeles, 2002)
- [Result] Baron-Cohen S, Jolliffe T, Mortimore C, Robertson M. Another advanced test of theory of mind: evidence from very high functioning adults with autism or asperger syndrome. J Child Psychol Psychiatry. 1997 Oct;38(7):813-22. doi: 10.1111/j.1469-7610.1997.tb01599.x. PMID 9363580
- [Result] Baron-Cohen S, Wheelwright S, Hill J, Raste Y, Plumb I. The "Reading the Mind in the Eyes" Test revised version: a study with normal adults, and adults with Asperger syndrome or high-functioning autism. J Child Psychol Psychiatry. 2001 Feb;42(2):241-51. PMID 11280420
- [Result] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Result] Wassermann EM, Grafman J, Berry C, Hollnagel C, Wild K, Clark K, Hallett M. Use and safety of a new repetitive transcranial magnetic stimulator. Electroencephalogr Clin Neurophysiol. 1996 Oct;101(5):412-7. PMID 8913194

RESULTS

PARTICIPANT FLOW:
Recruitment Details: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Groups:
- TMS and fMRI: * functional MRI
  * single and paired pulse TMS (to identify the difference of motor excitability between patients and healthy controls)
  TMS and functional MRI (Magstim): single and paired pulse low frequency TMS. 3T structural MRI scans, amplitude modulated continuous arterial spin labeling( CASL) perfusion imaging sequence optimized for 3T is employed for perfusion MR scans using GE FAIR sequence for parallel imaging.
Period: Overall Study
Arm/Group | TMS and fMRI
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Arm/Group | TMS and fMRI
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Gender
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Repetitive Behavior Scale-revised
Time Frame: during screening
Population: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Arm/Group | TMS and fMRI
Number analyzed (Participants) | 0

2. Secondary Outcome: Vineland Maladaptive Behavior Scale
Time Frame: during screening
Population: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Arm/Group | TMS and fMRI
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: P.I. has left the institution and NYSPI has no access to the data. Results will not be analyzed or presented.
Arm/Group | TMS and fMRI
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes